CLINICAL TRIAL: NCT01604330
Title: Alcohol Treatment: Pragmatic Therapeutic Trial Randomized, Double-blind for a Year in Ambulatory Care of Baclofen Versus Placebo.
Brief Title: Baclofen for the Treatment of Alcohol Drinkers
Acronym: BACLOVILLE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société de Formation Thérapeutique du Généraliste (Other); Cochin Hospital, Paris, Professor Claire Le Jeunne - Chief Scientist (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P110112; 2011-005787-17 (EudraCT Number)
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Alcoholism
Keywords: High dose baclofen; Alcoholism; Abstinence; Low risk consumption; Craving
MeSH Terms: conditions — Alcoholism | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Baclofen (Experimental): Baclofen will be administered orally for a maximum of 52 consecutive weeks. For the first 3 days, patients will receive baclofen in a dose of 5 milligrams three times a day; then the dose of baclofen will be increased to a maximum of 300 milligrams a day. In case of intolerance, dosage can be decreased.
  Interventions: Drug: Baclofen
- Placebo (Placebo Comparator): Sugar pill will be administered orally for a maximum of 52 consecutive weeks. For the first 3 days, patients will receive sugar pill in a dose of 5 milligrams three times a day; then the dose of sugar pill will be increased to a maximum of 300 milligrams a day. In case of intolerance, dosage can be decreased.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen — Baclofen will be administered orally for a maximum of 52 consecutive weeks. For the first 3 days, patients will receive baclofen in a dose of 5 milligrams three times a day; then the dose of baclofen will be increased to a maximum of 300 milligrams a day. In case of intolerance, dosage can be decreased.
  Arms: Baclofen
Drug: Placebo — Sugar pill will be administered orally for a maximum of 52 consecutive weeks. For the first 3 days, patients will receive sugar pill in a dose of 5 milligrams three times a day; then the dose of sugar pill will be increased to a maximum of 300 milligrams a day. In case of intolerance, dosage can be decreased.
  Arms: Placebo

SUMMARY:
The main objective of this study is to show the effectiveness to a year of baclofen compared to placebo, on the proportion of patients with a low risk alcohol consumption or no, according to the WHO standards.

DETAILED DESCRIPTION:
Baclofen, a gamma-aminobutyric acid 'B-receptor' agonist, has long been used to treat spasticity from neurological diseases, at a dose of 30-90 mg/day. It appears today to be a promising but controversial candidate for treating alcoholic patients (Enserick, 2011) by reducing or even suppressing their craving to drink. A few case reports (Ameisen, 2005; Bucknam, 2007; Dore et al., 2011) and a retrospective study (Rigal et al, 2012) suggest that some patients might respond favorably to baclofen at higher doses than 90 mg/day. This is a randomized controlled trial versus placebo testing such doses.

An extraction of patients DNA and a genetic analysis will be done after the end of the trial. In a gene candidate approach, the association of several genes with the efficiency of the treatment and its side effects, based on the literature, will be investigated using micro-array technology.

ELIGIBILITY:
Inclusion Criteria:

* Patient coming for a problem with alcohol (alcohol at high risk during the past three months (at least two times during each month) according to the WHO standards;. i.e.: in women more than 40 g per day or 280 g per week or more of 40 g at once; the man more than 60 g per day or 420 g per week or more than 60 g in once, and expressing the desire to be abstinent or to have a consumption to low level of risk).
* Volunteer to participate in the trial and having given his consent written after appropriate information
* Patient having no treatment for the maintenance of abstinence (acamprosate, naltrexone) and the prevention of relapse (disulfiram) for at least 15 days before the beginning of the trial
* Patient informed about the possibility of drowsiness in relation to the treatment and the associated risks to drive vehicles (motorized or not), the use of machines (including domestic use or recreation) and the execution of tasks requiring attention and precision
* Including woman of childbearing age (but taking effective contraception).

Exclusion Criteria:

* Patient taking already baclofen or having taken baclofen
* Patient pregnant, lactating, or childbearing years in the absence of effective contraception
* Patient with porphyria
* Patient with Parkinson's disease
* Patient with severe psychiatric pathology (psychosis, including schizophrenia and bipolar disorders) that can compromise the observance
* Patient with organic disease serious enough to not to allow its inclusion in the study according to the opinion of the investigator
* Patient homeless
* Patient without social cover
* Patient unable to properly follow-up book, cannot commit to one year of follow-up
* Patient with a contraindication to taking baclofen (intolerance to gluten by the presence of wheat starch
* Patient with a severe intolerance known about the lactose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2012-05-29 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Proportion of abstainer patients and patients with a low risk consumption | 12 months after the initiation of treatment
  Low risk consumption according to the criteria of WHO (World Health Organization). The assessment will be on the declarative of the patient (with autoquestionnaire). It will be compared between the two groups using a Chi-2 test.

SECONDARY OUTCOMES:
Distribution of Efficience dosage of baclofen | 12 months after the initiation of treatment
  Published studies indicate that the average dose would be about 140 mg per day without, a priori, report with the weight of the patient. Animal studies show an optimal dose of 3 mg/kg.
To evaluate the tolerance of baclofen | 12 months after the initiation of treatment
  To try, if possible, to differentiate which is due to the molecule, which is due to the stop of drinking alcohol and which is due to the alcohol-baclofen potentiation and looking for all the side effects including at high dosages.
To better characterize the alcoholic patients in whom this molecule is effective | 12 months after the initiation of treatment
  By using the anxiety/depression HAD scale. By using the scale of craving (Obsessive Compulsive Drinking Scale). By using the DSM - IV for the dependency.
Evolution of patients under treatment | 12 months after the initiation of treatment
  At each consultation, the consumption self-assessment questionnaire is analysed with the patient (book of follow-up) and missing data are sought and completed.
  To describe the evolution of patients under treatment from the point of view of the total consumption of alcohol, the monthly average consumption, the number of days of abstinence, the number of "heavy drinking days".
Cumulative quantity of alcohol drunk in the last month | 12 months after the initiation of treatment
  To analyse the cumulative quantity of alcohol drunk by the patient during the last month of treatment
Quality of life during treatment | at Day 1 and 12 months after the initiation of treatment
  To assess the quality of life during treatment by using the scale SF36 at the beginning and at the end of the study.
Evolution of biology | At day one, 6 months and 12 months after the initiation of treatment
  To study the evolution of biology, including liver, compared to the declaration made by the patient from his response to treatment. Biological examinations will be performed at the beginning, at 6 month and at the end of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jaury, MD, PhD, Principal Investigator — University of Paris 5 - Rene Descartes
Locations (1):
- Paris Descartes University, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rigal L, Sidorkiewicz S, Treluyer JM, Perrodeau E, Le Jeunne C, Porcher R, Jaury P. Titrated baclofen for high-risk alcohol consumption: a randomized placebo-controlled trial in out-patients with 1-year follow-up. Addiction. 2020 Jul;115(7):1265-1276. doi: 10.1111/add.14927. Epub 2020 Feb 16. PMID 31833590
- [Derived] Braillon A, Naudet F. Pharmacotherapies for Alcohol Use Disorder: Over Both Sides of the Atlantic Ocean. Mayo Clin Proc. 2020 Oct;95(10):2294-2295. doi: 10.1016/j.mayocp.2020.08.005. No abstract available. PMID 33012365